CLINICAL TRIAL: NCT04408768
Title: Stress Hyperglycemia as a Prognostic Factor in Acute Ischemic Stroke Patients
Brief Title: Stress Hyperglycemia and Acute Ischemic Stroke
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Hanaa Mohamed Abdallah ElGendy MD, Assistant Professor, Ain Shams University
Other Study IDs: El Zaiton Specialized Hospital
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2020-06-01 (Actual); Status verified 2020-05

CONDITIONS: Stress Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normal RBS: Normal RBS on ICU admission and controlled blood sugar within 24 hours
  Interventions: Other: standard protocol for stroke patients
- High RBS: High RBS on ICU admission and uncontrolled blood sugar during first 24 hours
  Interventions: Other: standard protocol for stroke patients

INTERVENTIONS:
Other: standard protocol for stroke patients — Standard protocol for stroke patients
  Other Names: no specific intervention

SUMMARY:
Whereas diabetes mellitus is clearly a risk factor for the occurrence of stroke and for its poor prognosis, hyperglycemia per se is also linked to increased morbidity and mortality in stroke patients.Therefore, the objective of this work was to study the glycemic status of acute ischemic stroke patients and to assess its impact on stroke outcome.

DETAILED DESCRIPTION:
Using PASS program, setting alpha error at 5% and power of 80%, the total sample size was estimated to be 80 cases.

The NIHSS was used as a primary outcome; 40 cases were needed in each group. Secondary outcomes were hemorrhagic transformation, hospital stay duration, mechanical ventilation, need for vasopressors, and 30-days mortality.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke within 24 hours of onset of symptoms

Exclusion Criteria:

* subdural hematoma
* Transient ischemic attack
* Subarachnoid hemorrhage
* Hemorrhagic stroke
* Major comorbidities Hyperglycemia on admission that was controlled (random blood sugar (RBS) < 150 mg/dl) within 24 hours with insulin therapy, diabetic
* Ketoacidosis
* RBS less than 70 mg/dl on admission

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included eighty acute ischemic stroke patients who presented within 24 hours of onset of symptoms. They were equally divided into two groups; group A included patients with normal (70-150 mg/dl) RBS on ICU admission and controlled blood sugar within 24 h, while group B included those with high RBS on ICU admission and uncontrolled blood sugar during first 24 h.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2019-07-09 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
National Institutes of Health Stroke Scale (NIHSS) | 30 days
  The NIHSS score categorized into: no stroke symptoms (0), mild stroke (1-4), moderate stroke (5-15), moderate to severe stroke (16-20), and sever (21-42)

SECONDARY OUTCOMES:
30-days mortality | 30 days
  Hemorrhagic transformation, the length of hospital stay, need for mechanical ventilation and vasopressors and 30-days mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Hanaa El Gendy, Cairo, Ain Shams University Specialized Hospital, Egypt

IPD SHARING:
Plan to Share IPD: Undecided